CLINICAL TRIAL: NCT05721222
Title: Phase 1/2 Study of PRO1160 in Patients With Metastatic Renal Cell Carcinoma (RCC), Metastatic or Relapsed Nasopharyngeal Carcinoma (NPC), or Advanced (Stage III or IV) Non-Hodgkin Lymphoma (NHL)
Brief Title: Trial of PRO1160 (GEN1160) in Relapsed or Refractory Non-Hodgkin Lymphoma (NHL) (PRO1160-001)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Genmab has decided to discontinue the clinical development of GEN1160 due to slow enrolment
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO1160-001 (GCT1160-01)
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Renal Cell Carcinoma; Nasopharyngeal Carcinoma; Non Hodgkin Lymphoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Nasopharyngeal Carcinoma; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GEN1160 (Experimental): GEN1160 monotherapy in escalating doses in the dose escalation part and at the recommended phase 2 dose in the expansion parts.
  Interventions: Biological: GEN1160

INTERVENTIONS:
Biological: GEN1160 — IV infusion of GEN1160
  Other Names: PRO1160

SUMMARY:
Brief Summary:

This study will test the safety, including side effects, and determine the characteristics of a drug called GEN1160 (PRO1160) in participants with solid tumors and blood cancers.

Participants will have cancer that has spread through the body (metastatic) or cannot be removed with surgery (unresectable) or relapsed or refractory to prior treatments.

This Phase 1/2 study will have three parts. The dose escalation part of the study will find out how much and how frequently GEN1160 should be given to participants. The expansion Part A and expansion Part B will use the dose and schedule found in the dose escalation part to find out how safe GEN1160 is and if it works to treat the diseases under study. The diseases under study will be Renal Cell Carcinoma (RCC), Nasopharyngeal Carcinoma (NPC) and Non-Hodgkin Lymphoma (NHL) in Escalation and diffuse large B-cell lymphoma (DLBCL) in expansion Part A and Part B.

DETAILED DESCRIPTION:
This is a Phase 1/2 study of GEN1160, a CD70 targeted antibody-drug conjugate, to evaluate the safety, tolerability, pharmacokinetics (PK), and antitumor activity of GEN1160 in participants with selected locally advanced /or metastatic solid and hematologic malignancies, including RCC, NPC and NHL. This study consists of 3 parts, Dose Escalation, Expansion Part A and Expansion Part B.

Dose escalation may evaluate up to 5 dose levels of GEN1160 on Day 1 of a 21 day cycle by intravenous (IV) infusion.

Expansion will be initiated at a dose level based on a comprehensive analysis of safety, tolerability, clinical PK, pharmacodynamics (PD) and activity data from the dose escalation. Expansion will be conducted in 1 cohort of up to 10 participants (expansion Part A) and 2 further cohorts (expansion Part B), each with up to 25 participants per cohort.

Participants will continue to receive study treatment until the first instance of disease progression, unacceptable toxicity, investigator decision, consent withdrawal, study termination by the Sponsor, initiation of non-GEN1160 anticancer therapy, participant noncompliance, pregnancy, or death.

ELIGIBILITY:
Dose Escalation: Key Inclusion Criteria:

* All participants must have pathologically confirmed diagnosis of one of the following tumor types:

  * Metastatic RCC, including clear cell renal cell carcinoma (ccRCC) or papillary RCC
  * Metastatic or relapsed Epstein Barr virus (EBV)-associated NPC not amenable to further local therapies (EBV association may have been determined by testing on tumor tissue or peripheral blood)
  * Advanced (Stage III or IV) NHL, including diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL) requiring systemic therapy, and mantle cell lymphoma (MCL)
* Participants must have relapsed or refractory disease following prior systemic therapies known to confer clinical benefit. At minimum, participants should have received the following therapies (unless deemed ineligible, refused by the participant, or not available in the region):

  * Participants with RCC must have received a minimum of one prior treatment regimen, and have received a tyrosine kinase inhibitor (TKI) and a programmed cell death (ligand) ([PD[L)])-1 inhibitor
  * Participants with EBV-associated NPC must have received a minimum of one prior treatment regimen, which must include a platinum-based chemotherapy regimen
  * Participants with DLBCL must have received a minimum of 2 prior treatment regimens, including a multi-agent chemoimmunotherapy regimen given with curative intent (eg, rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone [R-CHOP]), and participants must have received intensive salvage chemotherapy with hematopoietic stem cell transplant (HSCT) if considered eligible by the investigator
  * Participants with FL must have received a minimum of 2 prior treatment regimens, which must include a multi-agent chemoimmunotherapy regimen including an anti-CD20 agent
  * Participants with mantle cell lymphoma (MCL) must have received a minimum of 2 prior treatment regimens, which must include a multi-agent chemoimmunotherapy regimen including an anti-CD20 agent
* Measurable disease at baseline:

  * Participants with RCC and NPC must have measurable disease as defined per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 (Eisenhauer et al., 2009)
  * Participants with NHL must have measurable disease as defined by the Lugano Classification (Cheson et al., 2014)
  * Participants must be willing to provide a pre-treatment tumor specimen (archival or new tissue biopsy samples). If a new tissue biopsy is required, procedures more invasive than a core biopsy or significant risk procedures for which the procedure-associated absolute risk of mortality or major morbidity in the participant's clinical setting and specific institution is 2% or higher, should not be utilized.

Dose Escalation Key Exclusion Criteria:

* Prior treatment with anti-CD70 directed therapy
* Prior therapy with an antibody-drug conjugate (ADC) with a topoisomerase 1 inhibitor payload
* Prior allogeneic hematopoietic stem cell transplant (HSCT). Participants with prior autologous HSCT must have completed the procedure at least 100 days prior to the first dose of study drug.
* Known active central nervous system metastases, including carcinomatous meningitis. Participants with brain metastases may participate provided the metastases have been treated and are stable for at least 4 weeks prior to the first dose of study drug, they have no new or enlarging brain metastases and have discontinued corticosteroids prescribed for symptoms associated with brain metastases for at least 7 days prior to the first dose of study drug. Participants with a history of brain metastases, suspected new brain metastases, or a diagnosis of RCC should have a magnetic resonance imaging (MRI) of the brain at screening.

Expansion: Key Inclusion Criteria:

* Has pathological diagnosis of DLBCL, not otherwise specified (NOS) as defined by the World Health Organization (WHO) 2016 classification including both de novo or histologically transformed.
* Has relapsed or refractory disease with no available standard therapy or is not a candidate for available standard therapy, and for whom, in the opinion of the investigator, experimental therapy with GEN1160 may be beneficial. Participant must have received at least 2 systemic treatment regimens including CD20-containing chemoimmunotherapy.
* Has measurable disease according to the 2014 Lugano criteria (Cheson et al., 2014):

  * A fluorodeoxyglucose (FDG)-positron emission tomography (PET) scan demonstrating positive lesion compatible with computed tomography (CT)- or MRI-defined anatomical tumor sites; AND
  * A CT scan (or MRI) with involvement of ≥ 1 measurable nodal lesion (long axis > 1.5 centimeters (cm) and short axis > 1.0 cm) and/or ≥ 1 measurable extranodal lesion (long axis > 1.0 cm).
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Has a fresh biopsy (if clinically feasible and not considered as a high-risk procedure) or an archival tumor biopsy and submit to the central laboratory for CD70 assay
* Has acceptable laboratory test results per protocol

Expansion: Key Exclusion Criteria:

* Primary central nervous system (CNS) tumor or known CNS involvement.
* Has been exposed to any of the following prior therapies within the specified timeframes:

  * Received prior investigational CD70-targeting therapy, eg, CD70-directed chimeric antigen receptor T-cell (CAR-T) therapy, anti-CD70 monoclonal antibody (mAb), CD3 x CD70 bispecific monoclonal antibody (bsAb), or CD70 antibody-drug conjugate.
  * Autologous stem cell transplant within 60 days prior to the first dose of GEN1160.
  * Allogeneic stem cell transplant within 90 days prior to the first dose of GEN1160.
  * Chemotherapy within 2 weeks or major surgery within 4 weeks of the first dose of GEN1160.
  * Curative radiotherapy within 4 weeks or palliative radiotherapy within 2 weeks prior to the first dose of GEN1160.
  * Treatment with an investigational drug within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to the first dose of GEN1160 or currently receiving any other investigational agents.
  * Prior treatment with live, attenuated vaccines within 30 days prior to the first dose of GEN1160. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. Experimental and/or nonauthorized coronavirus disease (SARS-CoV-2) vaccinations are not allowed.
  * Receiving immunosuppressive drugs or systemic corticosteroids such as prednisone at doses > 25 milligrams (mg) daily or its equivalent within 14 days prior to the first dose of GEN1160.
* History of symptomatic autoimmune disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, Sjögren's syndrome, autoimmune vasculitis [eg, Wegener's granulomatosis]).
* Has clinically significant cardiac disease, including:

  * Myocardial infarction within 6 months prior to the first dose of GEN1160, or unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III or IV), cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE] Version 5.0 Grade 2 or higher), or clinically significant electrocardiogram (ECG) abnormalities.
  * Screening 12-lead ECG showing a baseline QT interval as corrected by QTcF > 480 milliseconds (msec).
  * Echocardiogram (ECHO) or multigated acquisition (MUGA) scan with left ventricular ejection fraction (LVEF) < 45%.
* Has clinically significant toxicities from previous anticancer therapies that have not resolved to baseline levels or to Grade 1 or lower. Note, participants with ≤ Grade 2 neuropathy or alopecia are an exception to this criterion and may qualify for the trial.
* Active graft versus host disease (GVHD) requiring immune suppression regardless of grade.

Note: Other protocol-defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to approximately 1 year
Dose Escalation: Number of Participants with Dose Limiting Toxicities (DLTs) | 28 days
Expansion Parts A and B: Objective Response Rate (ORR) | Up to approximately 1 year

SECONDARY OUTCOMES:
Dose Escalation: ORR | Up to approximately 1 year
Dose Escalation: Disease Control Rate (DCR) | Up to approximately 1 year
Dose Escalation and Expansion Parts A and B: Progression-free Survival (PFS) | Up to approximately 18 months
Dose Escalation and Expansion Parts A and B: Duration of Objective Response (DOR) | Up to approximately 1 year
Dose Escalation and Expansion Parts A and B: Peak Plasma Concentration (Cmax) of GEN1160-related Analytes | Up to approximately 1 year
Dose Escalation and Expansion Parts A and B: Time to Maximum Concentration (Tmax) of GEN1160-related Analytes | Up to approximately 1 year
Dose Escalation and Expansion Parts A and B: Area Under the Curve up to the Last Quantifiable Time-point (AUC0-last) of GEN1160-related Analytes | Up to approximately 1 year
Dose Escalation and Expansion Parts A and B: Number of Participants with Antidrug Antibodies (ADA) | Up to approximately 1 year
Expansion Parts A and B: Complete Response (CR) Rate | Up to approximately 1 year
Expansion Parts A and B: Overall Survival (OS) | Up to approximately 18 months
Expansion Parts A and B: Number of Participants with TEAEs | Up to approximately 1 year
Expansion Parts A and B: Number of Participants with Anti-GEN1160 Antibodies | Up to approximately 1 year
Expansion Parts A and B: Time-to response (TTR) | Up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (17):
- United States (14):
  - City of Hope Comprehensive Cancer Center - Duarte, Duarte, California
  - The City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Montefiore Medical Center - Montefiore Hospital, The Bronx, New York
  - Levine Cancer Center, Charlotte, North Carolina
  - Cleveland Clinic - Euclid Hospital, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Sarah Cannon Research Institute - Nashville, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - START Mountain Cancer Center, West Valley City, Utah
- China (3):
  - Cancer Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No